CLINICAL TRIAL: NCT03421366
Title: Modified Release Posaconazole in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 432.17
Record Dates: First submitted 2017-12-27; First posted 2018-02-05 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
Keywords: posaconazole
MeSH Terms: conditions — Cystic Fibrosis | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — As standard of care a pre-treatment sputum is collected for fungal cultures. The Aspergillus isolates collected will be retained and stored frozen for future testing of posaconazole susceptibility and whole genome sequencing to characterize clonal types and virulence properties
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cystic Fibrosis on Posaconazole: * Able to provide written informed consent
  * Greater than 18 years of age or older
  * Have a diagnosis of cystic fibrosis
  * No known azole hypersensitivity
  * To commence as part of their standard of care the newer modified release oral formulation of posaconazole to treat Aspergillus
  * Able to provide a pre-treatment sputum collected for fungal culture as part of standard of care
  * Have been prescribed a loading dose of 300mg bd for 1 day of the modified release posaconazole tablet followed by 300mg daily.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — A triazole antifungal drug that is used to treat invasive infections by Candida species and Aspergillus species in severely immunocompromised patients

SUMMARY:
A prospective single center observational cohort of patients with cystic fibrosis to determine whether adequate serum levels of posaconazole, after administration of the newer modified release once daily oral formulation, can be achieved.

DETAILED DESCRIPTION:
Use of antifungals has increased in people with cystic fibrosis. Aspergillus is the dominant fungal pathogen in this patient population and thus far, voriconazole has been used first line. Apart from recurrent and chronic lung infections, people with cystic fibrosis can also have problems with their gastrointestinal tract and absorption, and can develop chronic liver disease. As a consequence, they are at high-risk for not achieving adequate antifungal levels, which may be due to altered oral bioavailability, and they may be more susceptible to hepatic toxicities.

This study will evaluate the use of the newer modified release, once daily formulation of posaconazole in people with cystic fibrosis to identify if there is any difference in the bioavailability of the drug due to the effect of cystic fibrosis on the gastrointestinal tract. This newer formulation of once daily posaconazole is approved by the Therapeutic Goods Administration (TGA) and available on the Pharmaceutical Benefits Scheme (PBS) since March 2015. The newer formulation has the potential to overcome one of the major challenges with antifungals in cystic fibrosis; oral bioavailability. Posaconazole also appears to have reduced hepatotoxicity. This study will focus on the safety and tolerability of the drug, as well as pharmacological and microbiological endpoints.

20 eligible participants will be enrolled and have a

* Pre-treatment sputum will be collected as standard of care.
* Posaconazole serum levels will be taken at days 2, 5 and 7. (Day 5 and 7 as standard of care).
* renal and liver function assessed whilst on treatment as standard of care.
* followed up for 30 days to assess tolerability and monitor for the development of liver toxicity

ELIGIBILITY:
* Albe to provide written informed consent
* Greater than 18 years of age or older
* Have a diagnosis of cystic fibrosis
* To commence as part of their standard of care the newer modified release oral formulation of posaconazole to treat Aspergillus
* Able to provide a pre-treatment sputum collected for fungal culture as part of standard of care
* Have been prescribed a loading dose of 300mg bd for 1 day of the modified release posaconazole tablet followed by 300mg daily.

Exclusion Criteria:

* • Known azole hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cystic fibrosis attending care at the Alfred Hospital in Melbourne Australia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-02-05 (Estimated); Study Completion 2021-02-05 (Estimated)

PRIMARY OUTCOMES:
Serum levels of posaconazole in patients with cystic fibrosis taking the newer modified release once daily oral formulation. | 7 days
  Posaconazole serum levels at days 2, 5 and 7

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- See also: Rey E, Treluyer J, Pons G. Drug Dispostion in Cysytic Fibrosis. Clin Pharmacokinet 1998 Oct; 35 (4): 313-329 — https://link.springer.com/article/10.2165/00003088-199835040-00004